CLINICAL TRIAL: NCT00798473
Title: A Randomized Controlled Trial of Zoledronate in the Treatment of Osteopenia in Children and Adolescents With Crohn's Disease
Brief Title: Zoledronate for Osteopenia in Pediatric Crohn's
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Crohn's and Colitis Foundation (Other)
Responsible Party: Sylviane Forget, Assistant Professor of Pediatrics, McGill University Health Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCH002-56
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2008-11-26 (Estimated); Status verified 2008-11

CONDITIONS: Crohn's Disease; Osteopenia; Osteoporosis
Keywords: Crohn's disease; Osteopenia; Osteoporosis; Bisphosphonates; Zoledronate
MeSH Terms: conditions — Crohn Disease; Bone Diseases, Metabolic; Osteoporosis | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Zoledronic acid, 0.06 mg/kg IV in a single infusion, maximum of 4 mg
  Interventions: Drug: zoledronic acid
- 2 (Placebo Comparator): IV saline infusion
  Interventions: Other: IV saline infusion

INTERVENTIONS:
Drug: zoledronic acid — Zoledronic acid 0.066 mg/kg (maximum 4 mg) given as a single intravenous infusion over ten minutes
  Other Names: zoledronate; zometa
  Arms: 1
Other: IV saline infusion
  Arms: 2

SUMMARY:
Background:

* Up to 30% of children and adolescents with Crohn's disease have decreased bone strength, or decrease bone density, called osteopenia.
* Bisphosphonates are a group of drugs that have been well studied and found to be effective in the treatment of osteopenia in menopausal women.
* Zoledronate is a very potent third generation bisphosphonate, that is safe and easy to administer, and has been found effective in the treatment of menopausal women with osteopenia.

Hypothesis: The investigators hypothesize that zoledronate can improve bone density in children and adolescents with Crohn's disease with osteopenia.

DETAILED DESCRIPTION:
* This study is recruiting 40 children and adolescents, aged 6 to 18, who have a proven abnormal bone density as measured on a special type of x-ray called a DEXA-scan.
* Participants are allocated at random to one of two groups: either treatment with zoledronate, or a placebo.
* Neither the participants or the physicians are aware of which group each participant is in.
* Participants are followed every three months for one year, and assessed with blood tests, urine tests, physical examination, diet questionnaire and exercise questionnaire.
* Participants have a repeat DEXA scan at 6 and 12 months after beginning the study.
* Once all participants are enrolled and followed for one whole year, we will compare the bone density of the group treated with zoledronate with the group treated with placebo.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 6 to 18,
* diagnosed with Crohn's disease with osteopenia,
* a minimum of 6 months of adequate calcium and vitamin D intake. (Osteopenia was defined for the purposes of this study as: Z-score lumber spine BMD by DEXA of -2.0 or less, or -1.5 and a risk factor (either steroid use for 6 months or more or decrease of 0.5 z-score in the preceding 12 months).)

Exclusion Criteria:

* renal dysfunction,
* insufficient calcium or vitamin D intake,
* current medication or condition affecting bone metabolism,
* documented fracture, previously diagnosed bone disease,
* documented intolerance/hypersensitivity to bisphosphonates,
* previous treatment with bisphosphonates within the last 6 months.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2004-09; Primary Completion 2007-09 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Lumbar spine density by DEXA | 6 months

SECONDARY OUTCOMES:
Duration of effect by urinary bone metabolite markers | 6, 12 months
safety and tolerability (side-effects, renal and liver function, biochemical parameters) | 0, 3, 6, 12 months
Lumbar spine bone density | 12 months
Total body bone density | 12 months
Fractures | 0,3,6,12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sylviane Forget, MD MSc FRCPC, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Celia Rodd, MD FRCPC, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Center - Montreal Children's Hospital, Montreal, Quebec, Canada